CLINICAL TRIAL: NCT00891163
Title: A Randomized, Double-Blind, Two-Period, Crossover Study to Evaluate the Depth and Duration of Anesthesia of Synera™ Patches Compared to Placebo Patches Applied to Healthy Adult Volunteers
Brief Title: Evaluate the Depth and Duration of Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Senior Director, Clinical R&D, Endo Pharmaceuticals Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EN3274-101
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Pain
Keywords: Topical anesthesia; Analgesia
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synera (Experimental)
  Interventions: Drug: Synera™ Topical Patch (70 mg lidocaine/70 mg tetracaine)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: Synera™ Topical Patch (70 mg lidocaine/70 mg tetracaine) — 30 minute applicable on antecubital fossa
  Arms: Synera
Drug: Placebo Patch — placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the depth (mm) of anesthesia provided by the Synera topical patch (using sensory depth and pain depth evaluations), and to determine the duration (minutes) of anesthesia provided by the Synera topical patch (using dermal sensory testing and thermal sensory testing evaluations), compared with a matching heated placebo patch.

ELIGIBILITY:
Inclusion Criteria:

* Had no known significant diseases
* Normal 12-lead electrocardiogram
* Willing to refrain from using any local topical preparations

Exclusion Criteria:

* Taken over-the-counter (OTC) or prescription analgesics in any form within 24 hours
* Known allergy or sensitivity to any component of the Synera patch, including lidocaine, sympathomimetic amines, other local anesthetics of the amide type, epinephrine, or other patch components
* Had an active dermatological disease of any origin that may have interfered with their ability to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2006-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Sensory and pain depth measurements | 0, 30, 60, 90, 120 and 150 minutes
Dermal and thermal sensory testing evaluations | 0, 30, 60, 90, 120 and 150 minutes

SECONDARY OUTCOMES:
Assess the safety and tolerability of the Synera topical patch compared with a matching heated placebo patch | Throughout the study
Evaluate local effects on the skin at the site of patch application for dermal adverse events (AEs) | Throughout the study

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Medical Center, Thornton Hospital, San Diego, California, United States